CLINICAL TRIAL: NCT00389064
Title: A Multi-Centre, Double-Blind, Randomised, Parallel-Group, Placebo-Controlled Phase III Study of the Efficacy and Safety of Quetiapine Fumarate Sustained Release (Seroquel SR) in the Treatment of Elderly Patients With Generalised Anxiety Disorder
Brief Title: Efficacy and Safety Study of Seroquel SR in the Treatment of Generalised Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1448C00015; EUDRACT No: 2006-001195-21
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Results first posted 2009-06-23 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-03

CONDITIONS: Anxiety Disorders
Keywords: Generalised Anxiety Disorder; GAD
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Quetapine XR (Experimental): Tablets orally administered in flexible doses of 50 to 300 mg quetiapine XR once daily.
  Interventions: Drug: Quetiapine XR
- Placebo (Placebo Comparator): Matching placebo tablets orally administered once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine XR — Quetiapine XR 50 mg tablets orally administered in flexible doses of 50 to 300 mg quetiapine XR once daily, in the evening for a 9-week treatment period.
  Arms: Quetapine XR
Drug: Placebo — Matching placebo tablets orally administered in flexible doses of 50 to 300 mg once daily, in the evening for a 9-week treatment period.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate whether treatment with (SEROQUEL SR) quetiapine fumarate sustained release (SR) for 9 weeks compared to placebo will improve elderly patients with generalised anxiety disorder.

PLEASE NOTE: Seroquel SR and Seroquel extended release(XR) refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 66 years or older, with a documented clinical diagnosis of Generalised Anxiety Disorder (GAD).
* Absence of current episode of major depression.

Exclusion Criteria:

* The presence of dementia or other mental disorder than GAD.
* Serious suicidal risk, uncontrolled hypertension, substance or alcohol abuse.
* A current diagnosis of cancer or current or past diagnosis of stroke.

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 450 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Ruiz, MD, Study Director — AstraZeneca
Locations (43):
- United States (14):
  - Research Site, Fort Myers, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Miami, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Roswell, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Brooklyn, New York
  - Research Site, The Bronx, New York
  - Research Site, Avon Lake, Ohio
  - Research Site, Eugene, Oregon
  - Research Site, Jenkintown, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
- Estonia (3):
  - Research Site, Tartu, Estonia
  - Research Site, Tallinn
  - Research Site, Viljandi
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Gorlice
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Leszno
  - Research Site, Skorzewo
  - Research Site, Torun
  - Research Site, Wroclaw
- Russia (10):
  - Research Site, Arkhangelsk
  - Research Site, Izhevsk
  - Research Site, Lipetsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Stavropol
  - Research Site, Voronezh
- Ukraine (8):
  - Research Site, Hlevakha, Kyiv Oblast
  - Research Site, Dnipro
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kiev
  - Research Site, Luhansk
  - Research Site, Odesa
  - Research Site, Vinnitsa

REFERENCES:
- [Derived] Mezhebovsky I, Magi K, She F, Datto C, Eriksson H. Double-blind, randomized study of extended release quetiapine fumarate (quetiapine XR) monotherapy in older patients with generalized anxiety disorder. Int J Geriatr Psychiatry. 2013 Jun;28(6):615-25. doi: 10.1002/gps.3867. Epub 2012 Oct 16. PMID 23070803

RESULTS

PARTICIPANT FLOW:
Recruitment Details: International multi-center study, 47 sites recruited between Sept 2006 and Apr 2008
Pre-assignment Details: Screening for eligibility and wash-out of restriced medications
Groups:
- Quetiapine XR: Quetiapine fumerate XR - flexibly dosed (50 - 300 mg)
Period: Overall Study
Arm/Group | Quetiapine XR | Placebo
Started | 223 | 227
Completed | 178 | 168
Not Completed | 45 | 59
Not completed — Adverse Event | 11 | 3
Not completed — Lack of Efficacy | 3 | 14
Not completed — Withdrawal by Subject | 17 | 27
Not completed — Physician Decision | 2 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Multiple Reasons | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine XR | Placebo | Total
Number analyzed (Participants) | 223 | 227 | 450
Age, Customized [Number; unit: Participants]
  66 to 75 years | 197 | 195 | 392
  > 75 years | 26 | 32 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 157 | 318
  Male | 62 | 70 | 132

OUTCOME MEASURES:

1. Primary Outcome: Change in the Hamilton Rating Scale for Anxiety (HAM-A) Total Score
Description: HAM-A total score ( 0-56 units), 0 is the best, Change : score at week 9 minus score at randomization
Time Frame: Randomization to Week 9
Population: Modified Intent to Treat (MITT) population.
Measure: Least Squares Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 222 | 226
units on scale | -14.97 (7.4) [7.40 to 0.00] | -7.21 (7.8) [7.80 to 0.00]

2. Secondary Outcome: Change in Health-related Quality of Life as Measured by Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) Percent Maximum Total Score
Description: Q-LES-Q total score is the sum of the first 14 items of Q-LES-Q, and this total score is converted to a % maximum total score by : (Q-LES-Q total score -14) /56 x 100%, Larger values indicate a higher perceived quality of life enjoyment and satisfaction.
  Change : percentage at week 9 minus percentage at randomization
Time Frame: Randomization to Week 9
Population: In reporting Q-LES-Q there was missing data even with last observation carried forward (LOCF), so the total number of patients analyzed is 428 ( 211 Quetiapine XR and 217 Placebo).
Measure: Least Squares Mean (Standard Deviation); unit: Percentage of Maximum Total Score
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 211 | 217
Percentage of Maximum Total Score | 14.82 (12.40) [12.40 to 0.00] | 4.94 (11.60) [11.60 to 0.00]

3. Secondary Outcome: Change in the Clinical Global Impression - Severity of Illness (CGI-S) Score
Description: CGI-S score is accessed on a seven-graded scale ranging from most extremely ill/ very much worse (7) to normal/very much improved (1) , 1 is best Change : score at week 9 minus score at randomization
Time Frame: Randomization to Week 9
Population: Modified Intent to Treat (MITT) population.
Measure: Least Squares Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 222 | 226
units on scale | -1.76 (1.10) [1.10 to 0.00] | -0.59 (1.00) [1.00 to 0.00]

4. Secondary Outcome: Change in Psychic Anxiety Factor as Measured by HAM-A Psychic Cluster Score
Description: HAM-A psychic cluster score ( 0-28), 0 is the best Change : score at week 9 minus score at randomization
Time Frame: Randomization to Week 9
Population: Modified Intent to Treat (MITT) population.
Measure: Least Squares Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 222 | 226
units on scale | -8.88 (4.20) [4.20 to 0.00] | -3.81 (4.60) [4.60 to 0.00]

5. Secondary Outcome: Change in Somatic Symptoms as Measured by HAM-A Somatic Cluster Score
Description: HAM-A somatic cluster score (0-28), 0 is the best Change : score at week 9 minus score at randomization
Time Frame: Randomization to Week 9
Population: Modified Intent to Treat (MITT) population.
Measure: Least Squares Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 222 | 226
units on scale | -6.05 (4.00) [4.00 to 0.00] | -3.37 (3.90) [3.90 to 0.00]

6. Secondary Outcome: Hamilton Rating Scale for Anxiety (HAM-A) Response.
Description: HAM-A response, defined as 50% or greater reduction from randomization in HAM-A total score.
Time Frame: Week 9
Measure: Number; unit: Number of participants.
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 222 | 226
Number of participants. | 152 | 54

7. Secondary Outcome: Number of Patients Reaching Hamilton Rating Scale for Anxiety (HAM-A) Remission
Description: HAM-A remission, defined as HAM-A total score less or equal to 7. An indicator of HAM-A remission is calculated as:
  * If HAM-A total score≤7, THEN indicator=1
  * If HAM-A total score >7, THEN indicator=0
Time Frame: Week 9
Population: Modified Intent to Treat (MITT) population.
Measure: Number; unit: Number of participants.
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 222 | 226
Number of participants. | 89 | 29

8. Secondary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS)
Description: MADRS total score (0-60), 0 is best Change : score at week 9 minus score at randomization
Time Frame: Randomization to week 9
Population: Modified Intent to Treat (MITT) population.
Measure: Least Squares Mean (Standard Deviation); unit: units on scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 222 | 226
units on scale | -6.94 (4.70) [4.70 to 0.00] | -2.22 (4.70) [4.70 to 0.00]

9. Secondary Outcome: Change in the Visual Analogue Scale (VAS) Measuring Pain
Description: Visual Analogue Scale (VAS) measuring pain (0-100 mm), 0 is best Change : scale at week 9 minus scale at randomization
Time Frame: Randomization to week 9
Population: Modified Intent to Treat (MITT) population.
Measure: Least Squares Mean (Standard Deviation); unit: mm
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 222 | 226
mm | -17.95 (21.80) [21.80 to 0.00] | -6.18 (19.80) [19.80 to 0.00]

10. Secondary Outcome: Safety and Well Tolerated as Measured in Adverse Event
Description: Number of patients have at least one adverse event
Time Frame: From the start of treatment to last dose plus 30 days
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 223 | 227
Participants | 145.00 | 114.00

11. Secondary Outcome: Safety and Well Tolerated as Measured by Extra Pyramidal Symptoms (EPS)
Description: Number of patients have adverse events associated with EPS
Time Frame: From start of the study teatment to last dose plus 30 days
Population: Safety population
Measure: Number; unit: Patients
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 223 | 227
Patients | 12.00 | 5.00

ADVERSE EVENTS:
Arm/Group | Quetiapine XR | Placebo
Serious Adverse Events (participants affected / at risk) | 1/223 | 3/227
Other Adverse Events (participants affected / at risk) | 171/223 | 89/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR (N=223) | Placebo (N=227)
Bronchopneumonia (Infections and infestations) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR (N=223) | Placebo (N=227)
Dizziness (Nervous system disorders) | 30 | 16
Dry Mouth (Gastrointestinal disorders) | 37 | 16
Headache (Nervous system disorders) | 26 | 29
Nausea (Gastrointestinal disorders) | 20 | 9
Somnolence (Nervous system disorders) | 58 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to collaborate in good faith with AstraZeneca with regards to the contents and formation of any publication or disclosure to be made by the PI and to pay due consideration to the comments, views and opinions offered by AstraZeneca